CLINICAL TRIAL: NCT01947205
Title: Pain and Suction Curettage
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gökhan Açmaz (Other Government)
Responsible Party: Sponsor-Investigator, Gökhan Açmaz, Kayseri Education and Research Hospital, Kayseri Education and Research Hospital
Organization: Kayseri Education and Research Hospital (Other Government)
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Treatment
Other Study IDs: Kayseri ERH; KayseriERH (Other: KayseriERH)
Record Dates: First submitted 2013-09-16; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Curettage; Analgesia; Paracervical Block; Paracetamol
Keywords: Curettage; analgesia; paracervical block; paracetamol; lidocaine; Dexketoprofen trometamol
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen; dexketoprofen trometamol; Vacuum Curettage; Anesthesia, Obstetrical; Carticaine; Pharmaceutical Preparations

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- paracetamol (Active Comparator): Duration
  Interventions: Drug: paracetamol
- without drug (Active Comparator): Control group
  Interventions: Other: without drug
- dexketoprofen trometamol (Active Comparator): Study group
  Interventions: Drug: dexketoprofen trometamol
- two puff xylocain administration on cervical surface (Active Comparator): Study group
  Interventions: Drug: suction curettage
- paracervical block with ultracaine (Active Comparator): study group
  Interventions: Drug: suction curettage

INTERVENTIONS:
Drug: paracetamol
  Arms: paracetamol
Drug: dexketoprofen trometamol
  Arms: dexketoprofen trometamol
Drug: suction curettage
  Other Names: two puff xylocain administration
  Arms: two puff xylocain administration on cervical surface
Drug: suction curettage
  Other Names: paracervical block with ultracaine
  Arms: paracervical block with ultracaine
Other: without drug
  Arms: without drug

SUMMARY:
Aim of the study was to investigate the analgesic efficacy of preoperative oral dexketoprofen trometamol, intravenous paracetamol, lidocaine spray and paracervical block with ultracaine on curettage procedure.

ELIGIBILITY:
Inclusion Criteria:

* pregnant participants between 35-48 days of gestation (5 to 7 weeks of gestation) pregnant participants with a single viable intrauterine pregnancy requesting termination of pregnancy.

Exclusion Criteria:

incomplete abortions, diabetes mellitus, tendency to bleed such as thrombocytopenia, factor deficiency and functional disorders of platelets… etc, pelvic infection, known cervical stenosis, significantly impaired respiratory or cardiac conduction functions, active liver disease, renal disease, previous adverse reaction to any of the drugs used in the study, and patients who are unable to understand how to score a 10-cm visual analog scale (VAS) pain score. Moreover, patients who described chronic pelvic pain prior to the study or patients who rated their pain level on a continuous 100-mm VAS different from 0 (no pain) just before the study were not included into study.

Ages: 16 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 111 (Actual)
Dates: Start 2012-11; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
pain reduction | nine months

CONTACTS AND LOCATIONS:
Overall Officials: Gökhan Açmaz, MD, Principal Investigator — Kayseri Education and Research Hospital
Locations (1):
- Kayseri Education and Research Hospital of Medicine, Kayseri, Turkey (Türkiye)

REFERENCES:
- [Derived] Acmaz G, Aksoy H, Ozoglu N, Aksoy U, Albayrak E. Effect of paracetamol, dexketoprofen trometamol, lidocaine spray, and paracervical block application for pain relief during suction termination of first-trimester pregnancy. Biomed Res Int. 2013;2013:869275. doi: 10.1155/2013/869275. Epub 2013 Dec 24. PMID 24455735